CLINICAL TRIAL: NCT00980707
Title: Utility of Versican and Hyaluronan Measurement in Induced Sputum as Biomarker of Asthma
Brief Title: Utility of Versican and Hyaluronan Measurement in Induced Sputum as Biomarkers of Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Associated Scientists to Help Minimize Allergies (Other)
Collaborators: Benaroya Research Institute (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AI-005 versican
Record Dates: First submitted 2009-09-17; First posted 2009-09-21 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Allergic Asthma
Keywords: versican; hyaluronan; sputum
MeSH Terms: interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- inhaled corticosteroid (Experimental): All asthmatics will start inhaled corticosteroids.
  Interventions: Drug: Inhaled corticosteroid (fluticasone)

INTERVENTIONS:
Drug: Inhaled corticosteroid (fluticasone) — inhaled fluticasone 220 ug/bid
  Other Names: fluticasone

SUMMARY:
The purpose of this study is to determine the role of versican and hyaluronan measurements in induced sputum as biomarkers of asthma. Enroll 10 subjects with mild persistent asthma who are not receiving treatment with a controller therapy.

DETAILED DESCRIPTION:
We will compare spirometry, eNO and sputum measurements of versican and hyaluronan before and after treatment with fluticasone 220 ug/bid.

ELIGIBILITY:
Inclusion Criteria:

* Allergic asthma defined as a positive methacholine challenge

Exclusion Criteria:

* Non-atopic patients

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Compare hyaluronan and versican in asthmatics versus atopic non-asthmatics. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Leonard C Altman, MD, Principal Investigator — Associated Scientists to Help Minimize Allergies
Locations (1):
- Associated Scientists to Help Minimize Allergies, Seattle, Washington, United States